CLINICAL TRIAL: NCT02164214
Title: DOES ETANERCEPT INFLUENCE TWEAK MODULATION OF INFLAMMATION DURING INFLAMMATORY RHEUMATISMS (PSORIATIC ARTHRITIS AND RHEUMATOID ARTHRITIS)?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-002954-29; 2011-14 (Other: AP HM)
Record Dates: First submitted 2013-07-04; First posted 2014-06-16 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Inflammatory Rheumatism; Psoriatic Arthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Rheumatic Fever; Arthritis, Psoriatic; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients PSORIATIC ARTHRITIS (Experimental): etanercept Treatment
  Interventions: Drug: etanercept Treatment
- patients RHEUMATOID ARTHRITIS (Active Comparator): etanercept Treatment
  Interventions: Drug: etanercept Treatment

INTERVENTIONS:
Drug: etanercept Treatment

SUMMARY:
TWEAK (TNF weakly inducer of apoptosis) is a type II-transmembrane protein, member of the TNF ligand superfamily that can be cleaved to function as a soluble cytokine. Depending on target cell type, TWEAK triggers multiple cellular responses ranging from modulation of inflammation to cell death when it binds to its main receptor, Fn 14. Our team has been the first to describe pro-inflammatory effects of TWEAK during central nervous system inflammation. Various data support the possibility that TWEAK produced by synovial macrophages may contribute to chronic synovitis in animal models and in humans. In psoriatic arthritis (PsoA), anti-TNF therapy has been successful concording with the key role of TNF in the pathogenesis of this disease and the generation by psoriatic patients of neutralizing anti-TNF autoantibodies referred as "beneficial autoimmunity to pro-inflammatory mediators". In 2010, Van Kuijk et al. have described a high expression of TWEAK in the inflammatory synovial of PsoA and rheumatoid arthritis (RA) patients before and after anti-TNF therapy. The role of TNF-alpha in the regulation of TWEAK expression remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* · Group RhPso :
* Fill(Perform) the criteria CASPAR of the Rheumatism psoriasic (Taylor W, on 2006)
* rheumatoid Absence of factor and antibody anti-CCP(anti-post office account) (cyclic citrulline peptide) in the serum
* Indication established to begin a treatment with etanercept

  · Group PR
* Fill(Perform) the criteria of the ACR (American College of Rheumatology) for PR (revised in 1987) (Arneth FC, on 1988)
* Presence of antibody anti-CCP(anti-post office account) in the serum
* Indication established to begin a treatment with etanercept

Exclusion Criteria:

* Minors(Miners)
* pregnant or breast-feeding Women
* Adults under guardianship
* Nobody staying in a sanitary or social establishment
* Persons in emergency situation and/or not beneficiaries of a national insurance scheme
* Private persons of freedom
* Arthritis or not labelled polyarthritis
* Contraindication established in the treatment(processing) by etanercept
* PUVAthérapie or cyclosporine or high dose of corticosteroid therapy (except intra-articular infiltration) or other anti-TNF treatment(processing) in two months preceding the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
serum levels of soluble TWEAK | 42 months
  samples blood before and after etanercept Treatment

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Guis S, Berbis P, Stephan D, Bertin D, Amatore F, Balandraud N, Lesavre N, Desplat-Jego S. TWEAK-binding autoantibodies are generated during psoriatic arthritis and are not influenced by anti-TNF therapy. J Transl Med. 2016 Jun 23;14(1):185. doi: 10.1186/s12967-016-0923-8. PMID 27338143